CLINICAL TRIAL: NCT05072535
Title: A Single-dose, Randomized, Open-label, Two-period Crossover, Phase I Study to Evaluate Relative Bioavailability and Food-Effect of HA121-28 Tablet B in Healthy Subjects
Brief Title: A Study to Evaluate Relative Bioavailability and Food-Effect of HA121-28 Tablet B in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: HA122-CSP-005
Record Dates: First submitted 2021-09-28; First posted 2021-10-11 (Actual); Last update posted 2022-03-14 (Actual); Status verified 2021-11

CONDITIONS: Healthy Subjects

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part 1-Group A (Experimental): Subjects will receive 200 mg HA121-28 tablet A on Day 1 of the first cycle, followed by tablet B on Day 36 of the second cycle, in the fasted state.
  Interventions: Drug: HA121-28 tablet B; Drug: HA121-28 tablet A
- Part 1-Group B (Experimental): Subjects will receive 200 mg HA121-28 tablet B on Day 1 of the first cycle, followed by tablet A on Day 36 of the second cycle, in the fasted state.
  Interventions: Drug: HA121-28 tablet B; Drug: HA121-28 tablet A
- Part 2-Group C (Experimental): Subjects will receive 200 mg HA121-28 tablet B on Day1 of the first cycle in fasted state, followed by tablet B on Day 36 of the second cycle in the fed state.
  Interventions: Drug: HA121-28 tablet B
- Part 2-Group D (Experimental): Subjects will receive 200 mg HA121-28 tablet B on Day 1 of the first cycle in the fed state, followed by tablet B on Day 36 of the second cycle in fasted state.
  Interventions: Drug: HA121-28 tablet B

INTERVENTIONS:
Drug: HA121-28 tablet B — HA121-28 tablet B 200 mg
Drug: HA121-28 tablet A — HA121-28 tablet A 200 mg
  Arms: Part 1-Group A; Part 1-Group B

SUMMARY:
The study will be divided into 2 parts. The first part is a relative bioavailability study of HA121-28 tablet A and HA121-28 tablet B, and the second part is a food effect study of HA121-28 tablet B. Both Parts are single-dose, randomized, open-label, two-period crossover study to evaluate relative bioavailability HA121-28 tablet B in healthy subjects and the effect of food on pharmacokinetic profile of HA121-28 tablet B, respectively.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18 to 45 years (inclusive);
2. Body weight ≥ 50.0 kg (males) or 45.0 kg (females), body mass index (BMI) ranging from 18.0 to 26 kg/m^2 (inclusive);
3. Subjects who have normal or abnormal results without clinical significance after medical history, vital signs, 12-lead ECG, physical examination, laboratory tests (blood routine, blood biochemistry, coagulation function, urine routine, etc.) and other tests;
4. Subjects and their partners must take reliable non-hormonal contraceptive measures (such as condoms, non-drug intrauterine device, etc.) from signing informed consent until 6 months after study completion (except those who have taken permanent contraceptive measures, such as bilateral tubal ligation, vasectomy, etc.) and have no sperm or egg donation plan;
5. Be willing to sign an informed consent form (ICF) and complete the whole trial process according to the study protocol.

Exclusion Criteria:

1. Subjects with a previous history of allergy to 1 or more drugs or previous known other severe allergic reactions, including clear hypersensitivity to HA121-28 or equivalent and any excipients in this study, any food component;
2. Inability to swallow oral medications or presence of diseases that affect the safety evaluation and absorption, distribution, metabolism, or excretion of study medication;
3. Subjects with a clear history of neurological, or psychiatric disorder, or a history of serious cardiovascular, liver and kidney, endocrine, respiratory, blood, digestive and immune diseases, or a history of malignant tumour;
4. History of organic heart disease, heart failure, myocardial infarction, angina pectoris, unexplained cardiac arrhythmias, torsional ventricular tachycardia, ventricular tachycardia, QT prolongation syndrome or with symptoms of QT prolongation syndrome and family history (indicated by genetic proof or cardiac sudden death in a close relative at a young age);
5. Major surgery within 6 months prior to screening or planned surgery during the trial, including cosmetic, dental and oral surgery;
6. Subjects who had received the Novel Coronavirus vaccine within 1 month prior to screening;
7. Clinically significant ECG abnormalities: QTcF interval ≥450 ms (males) or 470 ms (females), or history of prolonged QTcF interval;
8. Any positive result for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab), human immunodeficiency virus antibody (HIV) or treponema pallidum antibody at screening;
9. Use of any prescription, over-the-counter (OTC), herbal medicine, nutritional supplements or health care products within 14 days prior to screening;
10. Regular consume of alcohol more than 14 units per week (One unit is equivalent to 285 mL beer, 25 mL spirits or 150 mL wine) within 4 weeks prior to screening, or a positive breath alcohol test at screening;
11. Subjects who smoke with an average of more than 5 cigarettes a day within 6 months prior to screening and unable to abstain during the study period;
12. Presence or history of drug abuse within 1 year prior to screening, or positive urine test for drug abuse at screening;
13. Habitual consumption of excessive drink or food containing caffeine or xanthine, such as coffee (>1100 mL per day), tea (>2200 mL per day), Cola (>2200 mL per day), energy drinks (>1100 mL per day), chocolate (> 510 g per day) within 4 weeks prior to screening, and subjects with special dietary requirements, not following the uniform diet;
14. History of needles or blood fainting, or have difficulty in blood collection;
15. Blood loss or donation more than 200 mL, or received blood transfusion within 4 weeks prior to screening, or plan on blood donation during the study period or within 1 month after the study;
16. Pregnant or lactating females;
17. Currently participating in other clinical studies, or participated in any clinical study and intake of study medication within 3 months prior to screening;
18. Not suitable for this study as judged by the investigator for any other reason.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-08 (Actual); Primary Completion 2021-12-19 (Actual); Study Completion 2022-03-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK) of HA121-28 in plasma: Area under the concentration-time Curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf). | predose (0)~288 hours post-dose
  AUCinf (unit: ng*h/mL)= Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf)
Pharmacokinetics (PK) of HA121-28 in plasma: Area under the concentration-time curve (AUC) from the time of dosing to the last measurable concentration (AUClast). | predose (0)~288 hours post-dose.
  AUC0-last(unit: ng*h/mL)=Area under the plasma concentration time-curve from zero to the last measured concentration
Pharmacokinetics (PK) of HA121-28 in plasma: Maximum concentration (Cmax) | predose (0)~288 hours post-dose.
  Cmax（ng/mL)=Maximum concentration

SECONDARY OUTCOMES:
Number of participants with Adverse Events (AEs) | up to Day 51.
  An AE is any untoward medical occurrence in a participant administered an IP, whether or not considered related to the IP. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of IP. This includes events related to the comparator and events related to the (study) procedures.
Number of participants with laboratory value abnormalities and/or adverse events (AEs) . | up to Day 51.
  Number of participants with potentially clinically significant laboratory values.
Number of participants with vital sign abnormalities and/or adverse events (AEs) . | up to Day 51.
  Number of participants with potentially clinically significant vital sign values.
Number of participants with electrocardiogram (ECG) abnormalities and/or Adverse Events (AEs) . | up to Day 51 .
  Number of participants with potentially clinically significant electrocardiogram (ECG) values.

CONTACTS AND LOCATIONS:
Locations (1):
- West China Hospital，Sichuan University, Chengdu, Sichuan, China